CLINICAL TRIAL: NCT03384186
Title: A Phase 1 Study to Evaluate the Pharmacokinetic Profile of ACH-0144471 Following Administration of Modified Release Prototype Formulations in Healthy Subjects
Brief Title: A Study of Modified Release Formulations of Danicopan in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ACH471-011; 2017-003525-15 (EudraCT Number)
Record Dates: First submitted 2017-12-14; First posted 2017-12-27 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: Danicopan; ALXN2040; ACH-0144471; Pharmacokinetics; Modified Release; Factor D Inhibitor; Relative Bioavailability
MeSH Terms: interventions — danicopan; rhoA GTP-Binding Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Danicopan Modified Release Prototype Tablets (Experimental): Participants received danicopan once each period as a single oral dose as follows:
  Period 1: Danicopan Modified Release Prototype 1 under fasted conditions. Period 2: Danicopan Modified Release Prototype 2 under fasted conditions. Period 3: Danicopan Modified Release Prototype 3 under fasted conditions. Period 4: Danicopan Modified Release Prototype 2 under fed conditions.
  There was a washout period of at least 14 days between each danicopan dosing.
  Interventions: Drug: Danicopan Modified Release Prototype 1; Drug: Danicopan Modified Release Prototype 2; Drug: Danicopan Modified Release Prototype 3

INTERVENTIONS:
Drug: Danicopan Modified Release Prototype 1 — Danicopan (400 milligrams [mg]) oral tablet.
  Other Names: ALXN2040; ACH-0144471 (formerly); ACH-4471; ACH4471; 4471
Drug: Danicopan Modified Release Prototype 2 — Danicopan (400 mg) oral tablet.
  Other Names: ALXN2040; ACH-0144471 (formerly); ACH-4471; ACH4471; 4471
Drug: Danicopan Modified Release Prototype 3 — Danicopan (800 mg) oral tablet.
  Other Names: ALXN2040; ACH-0144471 (formerly); ACH-4471; ACH4471; 4471

SUMMARY:
The purpose of this study was to evaluate and compare the plasma pharmacokinetic profiles of ACH-0144471 (danicopan) in healthy participants after administration of single oral doses of modified release prototype formulations.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18.0 to 30.0 kilograms/square meter.
* Female participants of childbearing potential must either agree to abstinence or use of a highly effective method of contraception.
* Male participants must either agree to abstinence or use of a condom plus an effective method of contraception.

Exclusion Criteria:

* Participants who have received any investigational medicinal product in a clinical research study within the previous 3 months.
* History of any drug or alcohol abuse in the past 2 years; current tobacco/nicotine user or within the last 12 months; positive drugs of abuse test result.
* Clinically significant laboratory abnormalities.
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder.
* History or family history of meningococcal infection.
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
* Presence or history of clinically significant allergy requiring treatment.
* Donation or loss of greater than 400 milliliters of blood within the previous 3 months.

Note: Other inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Time To Maximum Observed Concentration (Tmax) Of Danicopan After Treatment With Each Prototype Formulation | Up to 72 hours postdose
Maximum Observed Concentration (Cmax) Of Danicopan After Treatment With Each Prototype Formulation | Up to 72 hours postdose
Area Under The Concentration Versus Time Curve From Time 0 Extrapolated To Infinity (AUC0-inf) Of Danicopan After Treatment With Each Prototype Formulation | Up to 72 hours postdose

SECONDARY OUTCOMES:
Participants Experiencing Treatment-emergent Adverse Events | Day 1 (postdose) through follow-up visit (10 [+/- 2] days after last study drug administration)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes